CLINICAL TRIAL: NCT00191750
Title: Phase II Trial of ALIMTA in Relapsed Small Cell Lung Cancer
Brief Title: A Study of Pemetrexed in Small Cell Lung Cancer, Which Has Returned
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7209; H3E-US-S069
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Carcinoma, Small Cell
MeSH Terms: conditions — Carcinoma, Small Cell | interventions — Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed

SUMMARY:
The purposes of this study are to determine 1) the safety of pemetrexed and any side effects that might be associated with it 2) whether pemetrexed can help patients with small cell lung cancer live longer 3) whether pemetrexed can make tumors smaller or disappear and for how long and 4) to see if patients feel better while taking pemetrexed

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of small cell lung cancer
* One prior treatment with chemotherapy or immunotherapy with greater than 3 weeks since the prior treatment
* At least 18 years of age
* Estimated life expectancy of at least 12 weeks
* Ambulatory and capable of self-care(eg, up and about greater than 50% of waking hours)

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received FDA approval for any indication
* Less than 2 weeks from radiation therapy
* Other serious illness that would compromise the safety of the patient
* Most second primary malignancies treated less than 5 years previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-07; Study Completion 2006-09

PRIMARY OUTCOMES:
To assess the antitumor activity for patients with both sensitive and refractory small cell lung cancer patients as measured by tumor response rate. To characterize the toxicities of pemetrexed in this patient population

SECONDARY OUTCOMES:
To better understand any side effects of pemetrexed

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Dallas, Texas